CLINICAL TRIAL: NCT02880488
Title: Validation of a Questionnaire Assessing Quality of Life in Children With Amblyopia and Strabismus
Acronym: ASTEQ
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RBM_FAN_2013-7
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Amblyopia; Strabismus
MeSH Terms: conditions — Amblyopia; Strabismus

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
The validation of a French questionnaire is very important to assess rigorously and objectively the impact of the treatments of strabismus and amblyopia on children quality of life.

ELIGIBILITY:
Inclusion Criteria:

* children with a status of strabismus or not strabismus made by a specialized ophthalmologist
* children with a status of amblyopia or not amblyopia made by a specialized ophthalmologist
* signed consent of parents

Exclusion Criteria:

* ocular pathology (except for isolated ametropia)
* evolutive paralytic strabismus
* antecedent of surgery for strabismus
* strabismus surgery in the past 6 months
* disease with possible impact on the child's answers, such as severe neurologic troubles)
* poor knowledge of French language

Ages: 3 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Outpatients of pediatric ophthalmology will be included in the study. 50 patients will be included in each class of age: 3-4 years old; 5-7 years old; 8-17 years old.
  For each class of age, 50 children with strabismus or amblyopa will be included, half of which treated by eye occlusion ; and 50 children with no strabismus nor amblyopia, half of which wearing glasses.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
validation of the questionnaire | immediate

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France